CLINICAL TRIAL: NCT01617889
Title: Healthy Term Infants Fed Milk-Based Formulas With Different Fat Blends
Brief Title: Healthy Term Infants Fed Milk-Based Formulas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK88
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Term Infant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Powdered milk-based formula, standard fat blend (Active Comparator)
  Interventions: Other: A powdered milk-based infant formula, standard fat blend
- Powder milk-based formula, alternate fat blend (Experimental)
  Interventions: Other: Experimental powdered milk-based infant formula with an alternate fat blend

INTERVENTIONS:
Other: Experimental powdered milk-based infant formula with an alternate fat blend — formula to be consumed ad lib
  Arms: Powder milk-based formula, alternate fat blend
Other: A powdered milk-based infant formula, standard fat blend — formula to be consumed ad lib
  Arms: Powdered milk-based formula, standard fat blend

SUMMARY:
The objective is to assess the comparative fat and calcium absorption, and gastrointestinal (GI) tolerance in healthy normal term infants fed powdered milk-based formulas containing different fat blends.

ELIGIBILITY:
Inclusion Criteria:

* Infant is judged to be in good health.
* Infant is singleton from a full term birth
* Infant's birth weight was > 2490 g.
* Infant is between 53 and 115 days of age
* Infant is on infant formula and tolerating infant formula feedings
* Parent(s) confirm they will not administer vitamin or mineral supplements, solid foods or juices for the duration of the study, unless instructed otherwise by their healthcare professional.
* Parent(s) and physician agree to discontinue the use of medications or home remedies, herbal preparations that might affect GI tolerance

Exclusion Criteria:

Infant has received human milk within 7 days prior to SDay 1.

Any adverse maternal, fetal or infant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development and includes maternal substance abuse

Infant has been treated with antibiotics within 5 days prior to SDay 1

Infant has received probiotics within 5 days prior to SDay 1.

Ages: 53 Days to 115 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
calcium absorption | 8 days
  as measured in stool

SECONDARY OUTCOMES:
stool consistency | 28 days
  measured on 5 point scale
fat absorption | 8 days
  as measured in stool
average number of stools per day | 28 days
percent of feedings with spit up/vomit associated with feeding per day. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John Lasekan, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States